CLINICAL TRIAL: NCT00860483
Title: GAC 0201 Correlation of Laparoscopic Experience and Functional Brain Activation: A Pet Scan Study
Brief Title: Correlation of Laparoscopic Experience and Functional Brain Activation: A PET Scan Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Louis Kavoussi, Chairman of Urology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GCRC 0201
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Brain Function
Keywords: Comparison of experienced and novice laparoscopic surgeons
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- observational (No Intervention): This is an observational study. no intervention occurs in subjects. their performance in a laparoscopic trainer is observed and correlated with brain activity
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — PET Scan

SUMMARY:
The purpose of the research is to determine how practicing laparoscopic motor tasks affects the functional anatomy of the brain, and to investigate whether there is a correlation between surgical experience and functional brain activition. Additionaly, the investigators plan to use eye-tracking technology to see if the use of this technology can distinguish surgeons of various skill levels. The investigators hope that this study leads to new and effective methods of training surgical residents. All of the data will be collected at The Feinstein Institute for Medical Research, and may be used in future studies, which may or may not be related to urological diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Urology resident or fellow at Long-Island Jewish Hospital
2. Urology attending surgeon with previous laparoscopic experience
3. Medical Student Research Fellow with no previous laparoscopic experience
4. Right hand dominant subjects
5. No known neorologic defect reported by the subject -

Exclusion Criteria:

1. Left-hand dominant subjects
2. Self-reported neurologic defect reported by the subject -

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Laparoscopic experience | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Louis R. Kavoussi, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States